

### UVA CENTER FOR DIABETES TECHNOLOGY

# Evaluation of The Postprandial Impact of Automated Priming Bolus for Full Closed Loop Insulin Delivery

Protocol Chair

Sue A. Brown, MD

University of Virginia

Center for Diabetes Technology

NCT#05528770

Version Number: v1.7

06-Oct-2022



# **KEY ROLES**

| Protocol Principal Investigator | |
|---|---|
| Name, degree | Sue Brown, MD |
| Institution Name | University of Virginia Center for Diabetes Technology |



# PROTOCOL VERSION HISTORY

| Version<br>Number | Author(s) | Approver | Effective Date | Revision Description |
|---|---|---|---|---|
| 1.0 | Mark DeBoer,<br>Mary Oliveri | Sue Brown | 29-Jul-2022 | Original Protocol |
| 1.1 | Mary Oliveri | Mark DeBoer | 15-Aug-2022 | <ul> <li>FDA requested mods:</li> <li>Figure 1 was updated</li> <li>BPS transitions described (section 7.6)</li> </ul> |
| 1.2 | Mark DeBoer | Mark DeBoer | 16-Aug-2022 | <ul> <li>FDA requested mods:</li> <li>Inclusion &amp; exclusion criteria (section 3.5 &amp; 3.6)</li> <li>Pilot study BPS corrections (section 6.3 &amp; 6.4)</li> <li>Exercise termination criteria (section 7.8)</li> <li>Discharge criteria (section 7.9)</li> <li>Individual stopping criteria (section 11.10.1)</li> </ul> |
| 1.3 | Mary Oliveri | Sue Brown | 23-Aug-2022 | <ul> <li>FDA requested mods:</li> <li>Pilot study will complete a minimum of 2-3 participants (section 1.3, 3.2 &amp; Chapter 6)</li> <li>A H&amp;P within 9 months of screening appointments may be used (section 3.4 &amp; 3.7)</li> <li>Further modified Exercise termination criteria (section 7.8)</li> <li>Discharge criteria (section 6.6)</li> </ul> |
| 1.4 | Mary Oliveri | Sue Brown | 12-Sep-2022 | <ul> <li>IRB Pre-Review mods (07-Sep-2022):</li> <li>Clarified enrollment numbers (section 3.2 &amp; 13.2)</li> <li>Edited inclusion criteria (section 3.5).</li> <li>Edited Screening Process (section 3.4 &amp; 3.7)</li> <li>Deleted references to questionnaires (section 5.1, 7.2, &amp; 7.10)</li> <li>Added 5-minute low intensity warm up (section 7.7)</li> <li>Clarified Covid testing (section 9.1.3)</li> <li>Deleted Covid vaccination record (section 10.3)</li> </ul> |





| | | | | • Edited pre-screening description (section 3.7) |
|---|---|---|---|---|
| 1.5 | Sue Brown | Sue Brown | 25-Sep-2022 | <ul><li>IRB FB Review request:</li><li>SAP description (Chapter 13).</li></ul> |
| 1.6 | Mary Oliveri | Mary Oliveri | 27-Sep-2022 | IRB FB Review request: Remove screening remote references |
| 1.7 | Mary Oliveri | Mary Oliveri | 06-Oct-2022 | IRB FB Review request: |



#### SITE PRINCIPAL INVESTIGATOR STATEMENT OF COMPLIANCE

Protocol Title: Evaluation of The Postprandial Impact of Automated Priming Bolus for Full Closed Loop Insulin Delivery

Protocol Version/Date: v1.7 06-Oct-2022

I have read the protocol specified above. In my formal capacity as a Site Principal Investigator, my duties include ensuring the safety of the study participants enrolled under my supervision. It is understood that all information pertaining to the study will be held strictly confidential and that this confidentiality requirement applies to all study staff at this site.

This trial will be carried out in accordance with ICH E6 Good Clinical Practice (GCP) and as required by the following: United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 312, and/or 21 CFR Part 812).

As the Principal Investigator, I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the sponsor and documented approval from the Institutional Review Board (IRB), or other approved Ethics Committee, except where necessary to eliminate an immediate hazard(s) to the trial participants.

All key personnel (all individuals responsible for the design and conduct of this trial) have completed Human Participants Protection Training and Good Clinical Practice Training. Further, I agree to ensure that all staff members involved in the conduct of this study are informed about their obligations in meeting the above commitments.

| Investigator's Signature | Date: | / | / |
|-----------------------------------|-------|---|---|
| Investigator's Name: | | | |
| Site Name: University of Virginia | | | |



# LIST OF ABBREVIATIONS

| ABBREVIATION | DEFINITION |
|--------------|-------------------------------------------|
| ADRR | Average Daily Risk Range |
| AP | Artificial Pancreas |
| BG | Blood Glucose |
| BT/BTLE | Bluetooth, Bluetooth low energy |
| BPS | Bolus Priming System |
| CGM | Continuous Glucose Monitoring |
| CLC | Closed-Loop Control |
| CSII | Continuous Subcutaneous Insulin Injection |
| DKA | Diabetic Ketoacidosis |
| DSMB | Data Safety Monitoring Board |
| FCL | Fully Closed Loop |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HbA1c | Hemoglobin A1c |
| HBGI | High Blood Glucose Index |
| HIIT | High-intensity interval training |
| HCL | Hybrid Closed Loop |
| IDE | Investigational Device Exemption |
| IOB | Insulin-on-Board |
| LBGI | Low Blood Glucose Index |
| POC | Point-of-Care |
| QC | Quality Control |
| UI | User Interface |



# **PROTOCOL SUMMARY**

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| Title | Evaluation of The Postprandial Impact of Automated Priming Bolus for Full Closed Loop Insulin Delivery |
| Investigational Device | UVA Model Predictive Control Artificial Pancreas (RocketAP) with and without use of the Bolus Priming System (BPS) |
| Objectives | The purpose of this study is to show the safety and feasibility of a new fully automated AP controller with and without the Bolus Priming System |
| Study Design | A randomized cross-over trial assessing glycemic responses to a fully automated AP system using two approaches: |
| | 1) using the Bolus Priming System (which detects shifts in glucose level to trigger a priming dose of insulin) |
| | 2) without the Bolus Priming System |
| | We will also have structured meal and exercise challenges of the fully closed loop system. |
| Number of Sites | One |
| Endpoint | The primary outcome will be time in range 70-180 mg/dL for a 24-hour period. |
| Population | Key Inclusion Criteria |
| • | • Age 18 and ≤65 years of age |
| | • Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one |
| | year |
| | Currently using insulin for at least six months |
| | Currently using insulin pump for at least three months |
| Sample Size | • Pilot Study: complete a minimum of 2-3 participants |
| | Main Study: complete up to 20 participants |
| Treatment Groups | Randomized crossover: Participants will be randomized to the order that they experience |
| | the use of the BPS in fully automated closed loop (FCL) (for 24 hours each, with a 24-hour |
| | washout in between): 1) with the BPS active, 2) without BPS. <b>Pilot Study:</b> Participants will be admitted to a local hotel or rental house for up to |
| Participant Duration | approximately 24 hours and will have a dinner with the RocketAP without the BPS |
| | Main Study: Participants will be admitted to a local hotel for approximately 96 hours. |
| Due to cal Organian/Symonois | |
| Protocol Overview/Synopsis | Main Study participants will be admitted to the hotel for a 4-night study, receiving the two sessions in random order: 1) FCL with BPS activated, 2) FCL without the BPS, with a 24- |
| | hour washout period in between. During the admission, participants will receive structured |
| | meals and have blood glucose control followed to compare time in range 70-180 mg/dL |
| | between Controller sessions. After the first 24 hour period on the first FCL approach (BPS |
| | vs. no BPS,) that the participant has been randomized to, there will be a 24 hour challenge |
| | period before shifting to the other randomized approach; during this session participants will |
| | undergo further testing of the control algorithm, including meal challenges and a high- |
| | intensity interval training bout. |

### STUDY VISITS AND PROCEDURES SCHEDULE

| | Screening | Study Equipment<br>Training | Pre-Admission<br>Check-In | Study Admission | Post-Admission<br>Check-In |
|---|---|---|---|---|---|
| Location | Clinic | Clinic/ Remote | Phone/ Email/<br>Text | Hotel/Rental<br>House | Phone/ Email/<br>Text |
| Visit | 1 | 2 | 3 | 4 | 5 |
| Informed Consent | X | | | | |
| Eligibility Assessment | X | | | | |
| Medical History | X | | | | |
| HbA1c | X | | | | |
| Pregnancy test (if applicable) | X | X | | X | |
| Physical Exam | X | | | | |
| Vital Signs (height/weight) | X | | | X | |
| Electrocardiogram (ECG) | X | | | | |
| Demographic Survey | X | | | | |
| Randomization | | | | X | |
| COVID-19 Testing | | | X | | |
| CGM Use | | | | X | |
| Survey | X | | | | |
| Review diabetes management and AEs | | | | X | X |

Rocket-BPS 06-Oct-2022 

# TABLE OF CONTENTS

| 2 | Chapter 1 Background1 | 3 |
|----|---------------------------------------------------|---|
| 3 | 1.1 Introduction | 3 |
| 4 | 1.2 Study Objective | 4 |
| 5 | 1.3 Study Design 1 | 4 |
| 6 | 1.4 Study Device Download | 6 |
| 7 | 1.5 Study System Issues | 6 |
| 8 | Chapter 2 Study Devices1 | 8 |
| 9 | 2.1 Insulin Pump | 8 |
| 10 | 2.2 Continuous Glucose Monitor | 8 |
| 11 | 2.3 Blood Glucose Meter and Strips | 8 |
| 12 | 2.4 Ketone Meter and Strips | 8 |
| 13 | 2.5 Study Devices Accountability Procedures | 8 |
| 14 | Chapter 3 Study Screening1 | 9 |
| 15 | 3.1 Clinical Sites | 9 |
| 16 | 3.2 Participant Recruitment and Enrollment | 9 |
| 17 | 3.3 Informed Consent and Authorization Procedures | 9 |
| 18 | 3.4 Screening Procedures1 | 9 |
| 19 | 3.5 Participant Inclusion Criteria | 9 |
| 20 | 3.6 Participant Exclusion Criteria | 0 |
| 21 | 3.7 Visit 1: Screening Procedures | 1 |
| 22 | 3.8 Demographic Data Survey | 3 |
| 23 | Chapter 4 Randomization2 | 5 |
| 24 | 4.1 Pilot Study Participants | 5 |
| 25 | 4.2 Main Study Participants | 5 |
| 26 | Chapter 5 Visit 2: Study Equipment Training2 | 6 |

| 27 | 5.1 CGM Training | 26 |
|----|---------------------------------------------------|----|
| 28 | 5.2 Activity Tracker | 26 |
| 29 | 5.3 Study Insulin Pump | 27 |
| 30 | Chapter 6 Pilot Study | 28 |
| 31 | 6.1 Qualifications and Role of the Staff | 28 |
| 32 | 6.2 Visit 3: Pre-Admission Check-In Visit | 28 |
| 33 | 6.3 Visit 4: Admission Check-In | 28 |
| 34 | 6.4 Study Meals | 29 |
| 35 | 6.5 Admission Activities | 29 |
| 36 | 6.6 Admission Discharge | 29 |
| 37 | 6.7 Visit 5: Post Admission Check-In Visit | 30 |
| 38 | Chapter 7 Main Study | 31 |
| 39 | 7.1 Hotel Admission | 31 |
| 40 | 7.2 Qualifications and Role of the Staff | 31 |
| 41 | 7.3 Visit 3: Pre-Admission Check-In Visit | 31 |
| 42 | 7.4 Visit 4: Admission Check-In | 31 |
| 43 | 7.5 System Transitions | 32 |
| 44 | 7.6 Study Meals | 32 |
| 45 | 7.7 Admission Activities | 33 |
| 46 | 7.8 Admission Discharge | 34 |
| 47 | 7.9 Visit 5: Post Admission Check-In Visit | 34 |
| 48 | 7.10 Medical Monitor Review | 34 |
| 49 | Chapter 8 Medical Monitor Review | 35 |
| 50 | 8.1 Medical Monitor Study Safety Data Review | 35 |
| 51 | 8.2 Medical Monitor Main Study Safety Data Review | 35 |
| 52 | Chapter 9 Testing Procedures | 36 |
| 53 | 9.1 Laboratory / Point of Care Testing | 36 |

| 54 | Chapter 10 Risks Associated with Clinical Trial | 37 |
|----|-----------------------------------------------------------------|----|
| 55 | 10.1 Potential Risks and Benefits of the Investigational Device | 37 |
| 56 | 10.2 General Considerations | 40 |
| 57 | 10.3 COVID-19 Risk Mitigation Plan and Justification | 41 |
| 58 | Chapter 11 Adverse Events, Device Issues, and Stopping Rules | 42 |
| 59 | 11.1 Definitions | 42 |
| 60 | 11.2 Reportable Events | 43 |
| 61 | 11.3 Relationship of Adverse Event to Study Device | 44 |
| 62 | 11.4 COVID-19 Transmission | 44 |
| 63 | 11.5 Intensity of Adverse Event | 45 |
| 64 | 11.6 Coding of Adverse Events | 45 |
| 65 | 11.7 Outcome of Adverse Events | 45 |
| 66 | 11.8 Reportable Device Issues | 46 |
| 67 | 11.9 Timing of Event Reporting | 46 |
| 68 | 11.10 Stopping Criteria | 47 |
| 69 | 11.11 Independent Safety Oversight | 48 |
| 70 | 11.12 Definition of a Data Breach | 48 |
| 71 | Chapter 12 Miscellaneous Considerations | 49 |
| 72 | 12.1 Prohibited Medications, Treatments, and Procedures | 49 |
| 73 | 12.2 Participant Withdrawal | 49 |
| 74 | 12.3 Confidentiality | |
| 75 | Chapter 13 Statistical Consideration | 50 |
| 76 | 13.1 Design and Randomization | 50 |
| 77 | 13.2 Sample Size | 51 |
| 78 | 13.3 Outcome Measures | 51 |
| 79 | 13.4 Safety Analyses | 52 |
| 80 | 13.5 Baseline Descriptive Statistics | 52 |

| 13.6 Device Issues | 52 |
|---|---|
| Chapter 14 Data Collection and Monitoring | 53 |
| 14.1 Case Report Forms and Device Data | 53 |
| 14.2 Study Records Retention | 53 |
| 14.3 Protocol Deviations | 53 |
| Chapter 15 Ethics/Protection of Human Participants | 54 |
| 15.1 Ethics Standard | 54 |
| 15.2 Institutional Review Boards | 54 |
| 15.3 Informed Consent Process | 54 |
| Chapter 16 References | 56 |
| | Chapter 14 Data Collection and Monitoring |

92

# **Chapter 1 Background**

#### 1.1 Introduction

93

94

95

96

97

98 99

100

101

102103

104

105106

107

108

109

110111

A major impediment to maintaining blood glucose (BG) control in Type 1 diabetes (T1D) is missed meal boluses, which has been associated with significantly higher HbA1c levels. While the advent of the artificial pancreas (AP) offers promise of safe reductions in HbA1c, our research group previously found that current AP systems only partly compensates for missed prandial insulin.<sup>2</sup> We thus designed a new system called RocketAP to be fully automated, utilizing a Bolus Priming System (BPS) that recognizes meal ingestion and delivers a quick priming dose of insulin prior to extreme blood sugar excursions. When used as a fully automated closed loop (FCL) system (without any meal announcements to the controller), this system improves time-in-range compared to a current commercially available system (Control-IQ). However, we have not previously determined whether the BPS provides improved blood sugar control over what the RocketAP controller could without the BPS. Indeed, when the BPS provides a bolus, it reduces the amount of insulin the controller can provide in response to high blood sugars—leaving open the possibility that the RocketAP controller could provide a similar degree of blood sugar control after unannounced meals. In addition, this system needs to be further tested under challenging conditions of exercise and food intake. This is particularly true for the BPS, given the potential that the BPS could detect spurious changes in blood sugar and provide a priming dose of insulin in the absence of a meal.

- 112 In the current study, the maximum amount of insulin that the BPS injects (which varies based on
- the system's calculation of the probability that a meal has been ingested) is 6% of the person's
- total daily insulin for any individual meal. This system is equipped with a novel hypoglycemia
- anti-rebound system, which constrains insulin infusion after CGM/SMBG readings<70 mg/dL.
- The BPS system is also silenced at night (23:00 6:00h).
- 117 In the current study, we are testing this RocketAP system for BG levels using two approaches:
- 118 A randomized cross-over trial where each participant will experience FCL for two 24-hour study
- periods in random order (referred to as FCL1 and FCL2) with:
- The BPS functioning
- The BPS inactivated
- During the washout period between FCL1 and FCL2, we will test the RocketAP system in FCL
- 123 with further challenges, both before and after the change in BPS treatment arm—i.e., not as a
- 124 cross-over assessment but a comparison between participants randomized to start with or without
- 125 BPS. These challenges will include:
- A session of high-intensity interval training (assessing the safety of the BPS when BG's may spike during bursts of anaerobic activity)

Rocket-BPS 06-Oct-2022 

130

131

142

154

159

- A high-carbohydrate, high-fat meal (assessing how the system responds to prolonged carbohydrate absorption)
  - Ingestion of a bolus of simple sugar (assessing the safety of the BPS when the user's blood sugar spikes from a relatively low amount of carbohydrate)
- Participants will be admitted to a hotel and started on the RocketAP for the purpose of comparing
- FCL use with and without BPS as described above, all implemented on the DiAs platform (MAF
- 134 2109). As an assessment of the efficacy of the system in maintaining BG control, participants will
- be followed for approximately 24 hours in the randomized phase (FCL1 vs. FCL2) and during the
- 136 24-hour cross-over phase. Our primary outcome will be one of efficacy in assessing BG control
- 137 (TIR 70-180 mg/dL) between the two 24-hour FCL1/FCL2 periods.
- We hypothesize that performances of RocketAP without BPS in FCL will provide similar glycemic
- control as FCL with BPS. We expect that this will constitute an important step toward having a
- 140 fully automated AP system because it may remove the need for a BPS system that itself could
- increase risk of episodes of hypoglycemia.

### 1.2 Study Objective

- The purpose of this study is to test the performance of the RocketAP in FCL both with and without
- the BPS, assessing efficacy and safety. We will target completion of up to 20 adults in a
- randomized cross-over trial, comparing blood glucose time in range 70-180 mg/dL for two 24-
- hour periods and assessing TIR during an additional challenge period, which will be compared
- between those who started on BPS vs. those who did not.

### **1.3 Study Design**

- We will consent up to 30 participants, ages  $\ge 18.0$  and  $\le 65$  years, with a goal to have up to 20
- participants complete the trial. The study will be performed overnight at a local hotel/rental house
- 151 (heretofore referred to as "hotel"). Enrollment in the Pilot Study will proceed with the goal of
- 152 completing a minimum of 2-3 participants. This admission will be about 24 hours at a hotel/rented
- house. Enrollment in the Main Study will proceed with the goal of completing 20 participants.

#### 1.3.1 Study Hardware/Software

- 155 The study itself will involve use of the DiAs prototyping platform (MAF 2109), connected to a
- 156 Tandem t:AP research pump and a Dexcom G6 sensor, and implementing RocketAP with and
- without BPS. Upon arrival at the hotel, participants will be instructed in how to use the Tandem
- research pump as well as the UVa AP system, including stopping the system.

#### 1.3.2 Timing of UVa Artificial Pancreas Use

- 160 The participants will arrive to hotel the evening before starting the experimental system to allow
- for a settling of blood glucose in an unfamiliar environment. The next morning, participants will
- be connected to a Tandem research pump connected to the UVa DiAs platform and their Dexcom

Rocket-BPS 06-Oct-2022 

G6 Transmitter will be linked with DiAs. Participants will then be taught how to use DiAs in this configuration. The research pump will be programmed with the individual's usual insulin parameters. Once started, the participants will have their blood sugar managed through this system during the entirety of the time at hotel.

#### 1.3.3 Study Controller Sessions

Order and timing of controller sessions: During the hotel stay, participants will have two separate 24-hour periods during which they will receive FCL control with and without the BPS active. These will be separated by a 24-hour challenge period which will involve further challenges. The timing and potential order of these sessions is shown in Figure 1.



Figure 1: Timeline and randomized order of the Study Controller Sessions

During these 24-hour periods participants will be followed for the experimental meals as part of the Study Controller Sessions to compare blood glucose control with and without the BPS (Figure 1). The study meals and activities will be standardized between study sessions (see Figure 2).

Rocket-BPS 06-Oct-2022 

177178

179

180

181

182

183

184

185

186187

188 189

190

191

192

193

194

195

196

197

198

199

200

201

202

Figure 2: Timeline of Study Controller Sessions and Study Meals and activities. There will be two identical 24-hour periods (FCL1 in green and FCL2 in orange), separated by a 24-hour challenge period (FCL1 in green-hatched) that will first involve the BPS activation assignment the participant was randomized to (the treatment approach used in FCL1) and then involve the alternate assignment (the treatment approach to be used in FCL2), with the system switch at the end of the challenge day. Arrows represent meals with Blue Arrows representing meals in which the participants are using their personal devices.

The primary outcome will compare the percent time CGM is between 70 and 180 mg/dL during daytime for FCL1 and FCL2 sessions with and without BPS. During the time between arrival at the hotel and being started on the experimental system, participants will use their home diabetes management approach, including insulin dosing via normal carbohydrate announcement. Starting the first morning of the study (Day 2 of study), study staff who will be present will include nursing staff and technical staff; a study physician will be available either on-site or nearby off-site at all times. Hyperglycemia and hypoglycemia treatment protocols will be followed per guidelines. We anticipate more significant cases of hyperglycemia during meals on the study system because of the lack of carbohydrate announcement; participants will be encouraged to drink large amounts of non-caloric beverages, particularly after these meals. UVa CDT study staff will monitor CGM output continuously and manage glucose control issues. At the end of the hotel stay, the participant will return to their home insulin management.

#### 1.4 Study Device Download

Before discharge from the hotel, all study devices will be turned in to study staff for device download, and the participants will return to their usual diabetes management.

#### 1.5 Study System Issues

If the CGM signal becomes unavailable for more than 20 minutes consecutively, closed loop will not operate to automatically adjust insulin. If the CGM is not connected, the system will revert to usual function of the pump and deliver insulin with the insulin dosing parameters programmed in

Rocket-BPS 06-Oct-2022 

| 203 | the system for that individual. Resumption of closed-loop control will occur automatically once |
|---|---|
| 204 | CGM signal is available again. |
| 205 | If the study system is unable to maintain pump connectivity, the pump will automatically revert to |
| 206 | pre-programmed basal insulin delivery after 30 minutes without any need for instruction from the |
| 207 | user. |

Rocket-BPS 06-Oct-2022 

# **Chapter 2 Study Devices**

### **2.1 Insulin Pump**

- 210 The study systems will utilize the Tandem t:AP research pump connected to the UVa DiAs system
- 211 run on a dedicated external smart phone, running the RocketAP control algorithm with either the
- 212 BPS system active or not, with the order of these sessions determined randomly.

#### 2.2 Continuous Glucose Monitor

- The study CGM will include Dexcom G6 transmitter and sensors. The CGM sensor is viable for
- 215 10 days.

208

### 2.3 Blood Glucose Meter and Strips

- 217 Blood glucose levels will be measured during the hotel admission with the use of a study
- 218 glucometer. The CGM device will be calibrated, if needed, using the study glucometer and strips
- in accordance with the manufacturer's labelling.

#### 220 **2.4 Ketone Meter and Strips**

- 221 Blood ketone levels will be measured during the hotel admission with the use of the Abbott
- 222 Precision Xtra meters and strips in accordance with the manufacturer's labelling. The blood
- 223 glucose meter component of the Precision Xtra Device will not be used.

#### 2.5 Study Devices Accountability Procedures

Device serial numbers will be recorded, and use of equipment will be tracked.

### **Chapter 3 Study Screening**

#### 227 3.1 Clinical Sites

226

236

253

- The study will be performed at the University of Virginia, with screening procedures taking place
- either virtually, at the Clinical Research Unit, or at local hotel.

### 230 3.2 Participant Recruitment and Enrollment

- 231 Pilot Study: Enrollment goal in the Pilot Study will be to complete a minimum of 2-3 participants.
- Up to 6 participants may sign consent forms.
- 233 Main Study: Enrollment in the study will proceed with the goal of completing up to 20
- participants. Participants will initially be randomized for the order of using FCL with or without
- BPS. Up to 30 participants may sign the consent form.

#### 3.3 Informed Consent and Authorization Procedures

- 237 Before consent has been obtained, participants will be asked inclusion/exclusion criteria questions
- 238 during pre-screening to determine study eligibility. Before completing any procedures or
- collecting any data that are not part of usual care, written informed consent, when applicable) will
- be obtained. Potential eligibility may be assessed as part of a routine-care examination.
- 241 A participant is considered enrolled when the informed consent form has been signed by the
- participant and the study team.
- 243 Consenting procedures and documentation is defined in section 15.3.

#### 244 **3.4 Screening Procedures**

- 245 After informed consent has been signed, a potential participant will be evaluated for study
- eligibility through the elicitation of a medical history, performance of a physical examination
- by licensed personnel, an ECG, and pregnancy testing (if applicable) to screen for exclusionary
- 248 medical conditions.
- A physical exam documented in the prior 9 months can suffice for the physical exam but will not
- serve as an exclusionary criterion if not available. Participants may self-report height, weight,
- blood pressure, temperature, and heart rate. Individuals who do not initially meet study eligibility
- requirements may be rescreened at a later date per investigator discretion.

### 3.5 Participant Inclusion Criteria

- 254 The participants must meet all of the following inclusion criteria in order to be eligible to
- 255 participate in the study.
- 1. Age  $\geq$ 18.0 and  $\leq$ 65 years old at time of consent
- 257 2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year

- 258 3. Currently using insulin for at least six months
- 4. Currently using insulin pump for at least three months
- 5. Using insulin parameters such as carbohydrate ratio and correction factors consistently on their pump in order to dose insulin for meals or corrections
- 6. Current regular exercise (e.g. walk, bike, jog) and be able to participate in a high intensity interval training activity.
- 7. Access to internet and willingness to upload data during the study as needed
- 8. For females, not currently known to be pregnant or breastfeeding
- 9. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
- Willingness to suspend use of any personal CGM for the duration of the clinical trial once the
   study CGM is in use
- 273 11. Willingness to use the UVa closed-loop system throughout study admission
- 274 12. Willingness to use personal lispro (Humalog) or aspart (Novolog) during the study admission.
- 275 13. Willingness not to start any new non-insulin glucose-lowering agent during the course of the 276 trial (including metformin/biguanides, GLP-1 receptor agonists, pramlintide, DPP-4 277 inhibitors, sulfonylureas and naturaceuticals)
- 278 14. Willingness to eat at least 1 g/kg of carbohydrate per day during the hotel admission
- 279 15. Willingness to reschedule if placed on oral steroids
- 280 16. An understanding and willingness to follow the protocol and signed informed consent
- 281 17. Willingness to follow COVID-19 protocols in place at the time of study.

#### 282 **3.6 Participant Exclusion Criteria**

- The participant must not have any exclusion criteria in order to be eligible to participate in the study.
- 1. History of diabetic ketoacidosis (DKA) in the 6 months prior to enrollment
- 286 2. Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
- 288 3. Pregnancy or intent to become pregnant during the trial
- 4. Currently being treated for a seizure disorder
- 5. Planned surgery during study duration.
- 291 6. Treatment with meglitinides/sulfonylureas at the time of hotel study.

- 7. Use of metformin/biguanides, GLP-1 agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, or naturaceuticals with a change in dose in the past month.
- 8. Coronary artery disease or heart failure, unless written clearance is received from a cardiologist or personal health care provider allowing clearance for high-intensity interval training and documentation of a negative stress test within the year
- 9. History of cardiac arrhythmia (except for benign premature atrial contractions and benign premature ventricular contractions which are permitted or previous ablation of arrhythmia without recurrence which may be permitted)
- 300 10. Clinically significant electrocardiogram (ECG) at time of Screening, as interpreted by the study medical physician.
- 302 11. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:
  - a. Inpatient psychiatric treatment in the past 6 months
  - b. Presence of a known adrenal disorder
  - c. Abnormal liver function test results (Transaminase >2 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function
  - d. Uncontrolled thyroid disease
  - e. Musculoskeletal or other condition that limits participation in exercise portion of study
- 312 12. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.
- 314 13. Positive Covid-19 test result

304

305

306

307

308

309

310311

#### 3.7 Visit 1: Screening Procedures

- The participant will be evaluated for study inclusion and exclusion eligibility after the informed
- 317 consent form has been signed by the participant and the study team.
- Individuals who do not initially meet study eligibility requirements may be rescreened at a later
- 319 date per investigator discretion.
- 320 Screening procedures will last approximately 1-2 hours. The visit may occur in-person or by
- 321 telecommunication. The following procedures may be performed/data collected/eligibility criteria
- 322 checked and documented:
- 1. Inclusion and Exclusion criteria assessed
- 324 2. Demographics, including:
  - a. Date of birth
  - b. Gender
- c. Race

325

326

329

- d. Ethnicity
  - 3. Medical History, including diabetes history

Rocket-BPS 06-Oct-2022 

- 330 a. Duration of disease (number of years) b. Current insulin pump model 331 332 c. History of CGM use d. Current treatment 333 334 e. Severe hypoglycemia history f. Severe hyperglycemia history 335 g. History of seizures 336 h. Loss of consciousness 337 338 4. Basal rates 339 5. Carbohydrate ratios 340 6. Insulin sensitivity factors 7. Target glucose 341 342 8. Average daily insulin 343 9. Surgical history 10. Allergies 344 345 11. Concomitant medications 346 12. Electrocardiogram (ECG) 13. Physical Examination – Aa historical history and physical report within 9 months of 347 348 screening appointments may be used but is not required for eligibility. If vitals are not 349 available, may include self-reported values. 350 a. Weight (may be self-reported) b. Height (may be self-reported) 351 352 c. Blood pressure 353 d. Temperature 354 e. Heart Rate 355 14. Screening Labs a. Hemoglobin A1c point of care 356 357 b. Urine or serum pregnancy test for all women of childbearing potential (this test can 358 be done remotely with results sent to the study team) 359 If needed based on medical history, investigators may include baseline chemistry panel, liver function tests, hematocrit, and thyroid stimulating hormone (lab results within one year of 360 361 screening appointment may be used). 362 Up to 6 months of historical data from the participant's personal insulin pump, glucometer, or 363 continuous glucose monitor may be downloaded or recorded. Data will be obtained from the 364 participant's personal insulin pump and CGM. This data may be obtained through the commercial 365 applications (e.g. t:connect and Dexcom G6). 366 If participants are on-site, the participant's glucometer may be uploaded to ensure that the
- Any labs required may be obtained at a local laboratory (e.g. LabCorp) convenient to the

participant can successfully upload the equipment.

369 participant.

367

- This study is not meant to find out if the participant has any other disease or problem. The study
- leaders will alert the participant if any of the research results are important to his/her health during
- 372 the study. The participant may have a copy of the screening tests to discuss with the personal
- 373 physician. When the blood tests are completed, any blood left over will be thrown away. It will
- not be stored for any future testing.
- For potential subjects who live out of state and or a significant distance from UVA to facilitate the
- 376 consent process, e-consent will be used. Note: For potential participants who are not able to use
- DocuSign, email, fax, or mail will be an option for receipt of the signed consent. The consenting
- 378 process will involve discussing the study at length in a phone call/HIPAA compliant
- 379 telecommunication method with the interested potential participant. The potential participant will
- 380 be asked permission to review inclusion/exclusion criteria to assess if they are eligible to
- participate in the study. If permission is granted, the study team will review the pre-screening
- 382 questionnaire which contains the inclusion/exclusion criteria. If eligible, the study team member
- will provide a copy of the informed consent form (i.e. in person, email, or mail) to the potential
- participant for their review. Potential participants may also elect to choose to review the informed
- consent form prior to discussing pre-screening questions.
- The potential participant will be given an opportunity to ask the study team questions or may speak
- directly with the study physician. After ample time to make an informed decision, the potential
- participant may sign the consent form at home and provide it to the study team (e.g. in person,
- 389 electronically, email, fax, or mail). The potential participant's understanding of the information,
- presented in the process of consent will be assessed by asking open-ended questions, may occur
- during the phone call or at the screening appointment. Once consent is obtained, study procedures
- may begin (e.g. LabCorp).
- 393 The study physician or physician designee will have the discretion to repeat screening tests. The
- repeat screening tests may be conducted locally (e.g. LabCorp). The participant may request a
- 395 copy of any of the results from the screening evaluation to review with their primary care provider.
- 396 If an exclusionary condition is identified, the study participant will be excluded from participation
- with follow up and referral to their primary care physician as needed.
- 398 If the study participant is pregnant, the study physician will discuss the results of the blood test
- with the participant and the participant will be asked to seek confirmation of the test and the
- appropriate medical care.
- 401 Participants may be re-screened at a later date if their clinical situation changes as determined by
- 402 the study physician.

403

#### 3.8 Demographic Data Survey

Research in diabetes technology has revealed significant disparities in minoritized population's

405 representation in clinical trials and access to devices that improve diabetes outcomes. Collection

Rocket-BPS 06-Oct-2022 

406 of detailed demographic data regarding participants in technology trials has become essential. This includes data on race/ethnicity, income levels and insurance status, as well as education and other 407 variables that describe the study population. 408 The Demographic Data Survey will be electronically administered once eligibility has been met. 409 410 a. Gender 411 b. Race 412 c. Ethnicity d. Marital status 413 414 e. Level of education 415 f. Employment status g. Household income 416 417 h. Health insurance status 418 i. Monthly insulin costs

419

**Chapter 4 Randomization** 

| 420<br>421 | Participants will receive the two different experimental conditions (FCL with and without BPS) in random order as described below. |
|---|---|
| 422 | 4.1 Pilot Study Participants |
| 423 | Pilot participants will not be randomized and will use the RocketAP system with and without BPS. |
| 424 | 4.2 Main Study Participants |
| 425<br>426<br>427 | Once eligibility is met and screening procedures are completed, the participant may continue to randomization. Screening failures and study dropout participants may be replaced. Randomization will occur via permuted blocks of 4. |
| +∠ / | will occur via permitted blocks of 4. |

428

435

### **Chapter 5 Visit 2: Study Equipment Training**

- 429 Equipment training may begin at the hotel after UVa AP system has been put in place. The purpose
- of this training is to introduce the study insulin pump and study CGM to the participant.
- The participant's insulin parameters will be programmed into their study insulin pump and
- confirmed by two research staff. Subjects will then switch to the study insulin pump. The
- participant's personal pump and infusion site will be removed.
- The participant will have the insulin pump and sensor on them at all times.

#### 5.1 CGM Training

- 436 A study CGM will be provided to all participants at the training session. The participants will be
- provided with CGM equipment and instructed to use the study CGM on a daily basis. If the
- participant has prior use of the CGM, re-training will be specific to the individual. The study team
- 439 may elect to have less frequent CGM users watch the Dexcom online training videos
- 440 (https://www.dexcom.com/training-videos) to assist in the training session. Study staff training
- may include review of study CGM in real-time to make management decisions and how to review
- the data after an upload for retrospective review. Study staff will specifically identify how alarms
- are set using the app and the frequency that these alarms will repeat.
- The participants personal CGM will be discontinued. The participants will be observed placing the
- sensor and will learn/review how to access the CGM trace via the DiAs phone or the Tandem
- research pump, as needed. The participants will be asked to perform fingerstick blood glucose
- measurements (if needed) in accordance with the labelling of the study CGM device.
- An electronic copy of the CGM user's guide will be provided for the participants to read. The
- study team will be sure that the participants will leave the training session knowing how to properly
- use the CGM. The study team will be available for any questions.
- Participants will have the option of using their personal smartphone or receive a study smartphone
- 452 to use in order to collect the data from the devices. If the participant elects to use a personal device,
- 453 the Dexcom app will be downloaded to their phone in order to monitor the participant's CGM
- values and alerts in real-time may be used.

#### 5.2 Activity Tracker

- All participants may be asked to wear an activity tracker (e.g. Fitbit) during the entire study (home
- and hotel admissions) to record information about movement and heart rate though not an endpoint
- 458 in this study.

455

#### 459 5.3 Study Insulin Pump 460 The study team will be responsible for monitoring and managing the study insulin pump during the hotel admissions. The participants may be provided a quick overview on its functionality to 461 understand the equipment. 462 463 **5.3.1 Study Insulin Pump Topics** 464 The study team will assist the participant in study pump infusion site initiation and will start the 465 participant on the study pump. The study pump will be programmed with the participant's usual 466 basal rates and pump parameters. The participant's personal pump will be removed. The 467 investigator may elect to use an existing personal pump infusion site at their discretion at the start 468 of the study. 469 The participant will be instructed on charging the pump, navigation through menus, bolus 470 procedures including stopping a bolus, etc. 471 5.3.2 Other Issues The participant will be instructed to notify study staff if they experience any issues with the study 472 473 devices during the hotel admission. Staff will be present in the event that if insulin is delivered by 474 any means other than the study pump (e.g. injection of subcutaneous insulin via syringe in the 475 event of infusion site failure). If insulin is delivered by any means other than the study pump, the 476 study team will be instructed to turn off closed-loop mode for approximately four hours. 477 The participant will also be asked to alert the study clinical staff for technical issues with the 478 Tandem research pump and/or the DiAs system, including use of the study pump and study CGM 479 (open loop mode) during periods of component disconnections or technical difficulties. 480 A glucagon emergency kit will be available at the hotel once the investigational system is in place. 481 Glycemic Treatment Guidelines will be available for staff use during the study admissions. 482 **5.3.3 Optimization of Insulin Pump Settings** 483 Data-driven optimization of pump settings can occur any time prior to the hotel admission, 484 particularly if the participant contacts the study physician due to concerns about their pump 485 settings due to recurring hypo- or hyperglycemia. No pump settings changes can occur during 486 closed loop testing.

### **Chapter 6 Pilot Study**

- In order to optimize the flow of the study visits during the Main Study, we will perform a Pilot
- Study at a local hotel or rental house. The duration of the pilot admission will be approximately
- 490 24 hours with the intent of testing the logistics of our study procedures. The goal will be to
- complete 2-3 participants. Pilot study participants are eligible to enroll in the Main Study.
- 492 Participants and staff will adhere to the Covid-19 Mitigation Plan as outlined in Section 10.3

#### 6.1 Qualifications and Role of the Staff

- For the pilot study, there will be at least two study staff present at all times at the study site, at least
- one of whom will be clinical staff (e.g. nurse, physician, nurse practitioner, physician assistant).
- There will be a physician available either on-site or off-site within an approximate 20-minute drive
- at all times. In addition, one of the study medical physicians and one senior engineer will be on
- 498 call during the entire admission. Glucagon for the emergency treatment of hypoglycemia will be
- available on-site.

487

493

500

503

504

505

506507

508

509

510511

512

#### 6.2 Visit 3: Pre-Admission Check-In Visit

- Pilot participants will be contacted by the study team approximately 24-48 hours prior to the hotel admission to verify the following information:
  - Inquire about any changes to the participant's medical history
    - Study equipment (e.g. CGM and activity tracker) initiation has occurred
    - Determine pump profile(s) the participant uses on certain days
  - New CGM sensor has been placed approximately 24-72 hours prior to admission for proper warm-up
    - Verify with the participant that the goal CGM reading on day 2 is less than 200 mg/dL; this may require contact with the study physician prior today 2 of the hotel study.
    - Should any concerns regarding medical history, pump information, or unforeseen issues arise, the admission will be cancelled for that participant at the discretion of the investigator

#### 6.3 Visit 4: Admission Check-In

- 513 For the pilot study, one to three participants will be assessed at a time. The participant will arrive
- at the hotel on the first day of the admission. The study team will perform vital signs and inquire
- about any changes to the participant's medical history. Any changes to medical history will be
- 516 communicated to the medical physician to ensure continued eligibility and participation.
- A urine pregnancy test will be collected if relevant. The test must be negative for the participant
- 518 to continue with the study.
- The subject's CGM reading, and ketone concentration will be recorded. In the event that the
- 520 participant's CGM reading is not between 80-250 mg/dL or ketone concentration is ≥0.6 mmol/L
- 521 prior to initiation of the UVa AP system, the study physician may recommend additional insulin

- dosing according to the participants' usual doses. Study physician may elect to cancel participant's
- 523 participation in the hotel admission if concerned about their medical safety. This participant will
- 524 not be replaced.
- The participant's home insulin pump will be discontinued, and the study Tandem research insulin
- 526 pump will be initiated using the RocketAP system with BPS activated. The study team will ensure
- 527 the proper function of the CGM, insulin pump, and activity tracker. The goal will be to initiate
- 528 Closed-Loop Control by approximately lunch time, running the RocketAP system on the DiAs
- 529 platform.
- 530 The CGM used in the study is FDA-approved for the non-adjunctive measurement of blood
- glucose (i.e. the CGM reading can be used for insulin dosing decisions). The CGM readings will
- be the primary source of blood glucose values. There are no protocol fingerstick blood glucose
- measurements other than at times of CGM calibration (if necessary) and if directed by the study
- team. Fingerstick blood glucose measurements may be taken whenever participants experience
- symptoms, if the CGM glucose is suspected to be erroneous, or any time the participant would like
- 536 to be reassured.

537

542

### 6.4 Study Meals

- Participants will eat a structured dinner at approximately 6-7 pm during the admission. The
- participant will not announce carbohydrate ingestion, allowing testing of the RocketAP controller
- 540 with BPS following dinner. Breakfast in the morning will be with the BPS system engaged.
- Throughout the Pilot study, the participant will remain in closed loop mode.

#### 6.5 Admission Activities

- In the afternoon after admission, participants will participate in a supervised bout of high-intensity
- interval training (see details in Section 7.8). During this time, the system will have BPS activated.
- 545 Apart from the programmed exercise portions, participants will be free to engage in low-intensity
- activity (i.e. walking) during the admission. Participants will enjoy quiet activities in the evening.

#### 547 **6.6 Admission Discharge**

- 548 Discharge will be at approximately noon. Discharge criteria is CGM value 80-300 mg/dL with
- stable trend and ketones <=0.6 mmol/L. If the CGM values are above 300 mg/dL and ketone values
- are >0.6 mmol/L, the study team will check the insulin pump infusion site and correction insulin
- will be administered per study physician judgement via the subject's insulin pump. A qualified
- clinical study team member (e.g. MD, NP, PA, CDE) will assess and discuss the transition back to
- usual care with the study participant.
- Participants will be asked to continue monitoring ketone levels for 24-48 hours after the hotel
- admission if ketones were >0.6 mmol/L at time of discharge. Urine ketone supplies may be
- provided for this testing.

Rocket-BPS 06-Oct-2022 

### 557 **6.7 Visit 5: Post Admission Check-In Visit**

Approximately 24-48 hours after the hotel admission, the study team will contact the participant via phone/email/text/text to assess adverse events, adverse device effects, and device issues.

Rocket-BPS 06-Oct-2022 

# **Chapter 7 Main Study**

#### 7.1 Hotel Admission

560

561

565

577

581

582

583584

585

586

587

588

589

590

591

- Main Study participants will participate in hotel admission. Each admission will be up to
- approximately 96 hours in duration.
- Participants and staff will adhere to the Covid-19 Mitigation Plan as outlined in Section 10.3.

### 7.2 Qualifications and Role of the Staff

- There will be at least two study staff present at all times at the study site, at least one of whom will
- be clinical staff (e.g. nurse, physician, nurse practitioner, physician assistant). There will be a
- 568 physician at the hotel or nearby on call during the study at all times. In addition, at least one senior
- engineer will be on call during the entire admission. Participants will be remotely monitored by at
- 570 least one study team member using a web-based remote monitoring system that has been
- 571 previously established for DiAs. The web-based remote monitoring system will display real-time
- insulin delivery, CGM and other system information to allow for patient safety monitoring. In
- addition, study team members will be trained in all protocol and glycemic treatment guideline
- 574 procedures. The closed-loop system will be managed by the participant with study-staff
- supervision, particularly at the time of insulin boluses. Glucagon for the emergency treatment of
- 576 hypoglycemia will be available on-site.

#### 7.3 Visit 3: Pre-Admission Check-In Visit

- Participants will be contacted by the study team approximately 24-48 hours prior to each hotel
- admission if most recent contact with the study participant exceeds 10 days. The study team will
- verify the following information:
  - Inquire about any changes to the participant's medical history
    - Study equipment (e.g. CGM and activity tracker) initiation has occurred
    - Determine pump profile(s) the participant uses on certain days
    - New CGM sensor has been placed approximately 24-72 hours prior to admission for proper warm-up
    - Verify with the subject that the goal CGM reading at time of arrival is less than 200 mg/dL;
       this may require contact with the study physician prior to arrival on the day of the study visit
    - Should any concerns regarding medical history, pump information, or unforeseen issues arise, the admission will be cancelled for that participant at the discretion of the investigator

#### 7.4 Visit 4: Admission Check-In

- Participants will arrive at the hotel on the first day of the admission. As described in section 10.3,
- all participants will receive a test for COVID-19 after arriving for the study. The study team will
- 594 perform vital signs and inquire about any changes to the participant's medical history. Any

Rocket-BPS 06-Oct-2022 

- changes to medical history will be communicated to the medical physician to ensure continued
- eligibility and participation.
- A urine pregnancy test will be collected for female participants of childbearing age. The test must
- be negative for the participant to continue with the study.
- The subject's CGM reading, and ketone concentration will be recorded. In the event that the
- participant's CGM reading is not between 80-250 mg/dL or ketone concentration is ≥0.6 mmol/L
- prior to initiation of the UVa artificial pancreas system, the study physician may recommend
- additional insulin dosing according to the participants' usual doses. Study physician may elect to
- cancel participant's participation in the hotel admission if concerned about their medical safety.
- This participant will not be replaced.
- The participant's home insulin pump will be discontinued, and the study insulin pump will be
- 606 initiated. The study team will ensure the proper function of the CGM, insulin pump, and activity
- 607 tracker.

616

626

- The CGM used in the study is FDA-approved for the non-adjunctive measurement of blood
- glucose (i.e. the CGM reading can be used for insulin dosing decisions). The CGM readings will
- be the primary source of blood glucose values. There are no protocol fingerstick blood glucose
- 611 measurements other than at times of CGM calibration (if necessary) and if directed by the study
- 612 team. Fingerstick blood glucose measurements may be taken whenever participants experience
- symptoms, if the CGM glucose is suspected to be erroneous, or any time the participant would like
- to be reassured. Glycemic Treatment Guidelines to be used during the hotel admission are defined
- in a separate document.

#### 7.5 System Transitions

- Participants will be informed beforehand and at the time of the transfer from one BPS state to
- another. Participants will be told what this transition means with respect to insulin dosing. The
- transfer from one treatment to another will proceed as follows:
- The system is stopped
- DiAs is plugged into a laptop and 'parameters.xml' file (with the corresponding BPS
- 622 condition) will be replaced
- DiAs is restarted
- CGM is recovered and pump connections is checked
- DiAs is transitioned to Closed Loop Control mode

#### 7.6 Study Meals

- Participants will eat structured study meals during the admission, with the same amount of
- 628 carbohydrate, protein and fat for meals (breakfast, lunch, dinner) on the days for FCL1 and FCL2).
- During the 24-hour challenge period, there will be additional meal challenges that will only be
- performed on that day. This includes a high carbohydrate high fat meal at dinner (such as pizza)

and an early breakfast that consists primarily of fast-acting carbs (e.g., juice). In all cases the carbohydrate content of the meal will not be announced during the study once the AP system has been placed. Snacks with carbohydrates will not be allowed unless for the treatment of low blood sugars. Non-carbohydrates snacks may be allowed throughout the protocol per investigator discretion, but the intention is not to have non-carbohydrate snacks. Blood glucose levels will be followed via continuous glucose monitor and glucose values will be managed by the AP system as usual.

#### 7.7 Admission Activities

638

- During the study, we will challenge the participants with exercise sessions that will be supervised by study staff. During FCL1 and FCL2, participants will do a mild to moderate walking or similar exercise at approximately 4pm on each of those study days.
- 642 During the challenge phase (the 24-hour period between the FCL1 and FCL2), participants will 643 undergo supervised session of high-intensity interval training (HIIT). The HIIT workout will 644 consist of a 5-minute low intensity warmup period, a workout of about 1 minute of vigorous 645 exercise followed by approximately 2 minutes of light intensity exercise or rest. This 3-minute set 646 of intervals may be repeated up to 6 times or until volitional exhaustion, followed by approximately 647 5 minutes of light intensity cooldown and stretching. The goal of this will be to assess the safety of the AP system in HIIT, given that HIIT has been observed to result in an increase in BG levels, 648 649 which could theoretically lead to activation of the BPS—dosing insulin. The AP system will be monitored for BPS activation during this workout. If the BPS is activated, participants will 650 651 continue to be monitored for BG excursions, including receiving treatment for hypoglycemia if 652 this occurs (as described in the Glycemic Treatment Guidelines).
- Exercise challenges will be terminated early with subjective symptoms such as shortness of breath, chest pain, dizziness, palpitations, or any such concerning symptoms reported by participants. Participants will stop their participation in the exercise portion of the study if reporting any concerning symptoms. Study physicians (or physician's assistants) will assess the participants for their need for additional care outside the study. If symptoms resolve entirely and there is no additional requirement for care outside the study, participants will stop participation in the exercise portion of the study and will not repeat that portion of the study. Participants however may then
- 660 continue with the remainder of the study per investigator discretion.
- Participants will also be free to engage in low-intensity activity (i.e. walking) during the hotel
- admission but will be asked to have this match between 24-hour study periods as best as possible.
- Participants may leave the hotel to be outside, provided they are accompanied by a study staff
- member and follow COVID precautions in place at the time of study, as described in Section .3.
- Participants will enjoy quiet activities in the evening.

Rocket-BPS 06-Oct-2022 

| 666 | 7.8 Admission Discharge |
|---|---|
| 667<br>668<br>669<br>670<br>671<br>672 | Discharge will be at approximately 1 pm. Discharge criteria is CGM value 80-300 mg/dL with stable trend and ketones <=0.6 mmol/L. If the CGM values are above 300 mg/dL and ketone values are >0.6 mmol/L, the study team will check the insulin pump infusion site and correction insulin will be administered per study physician judgement via the subject's insulin pump. A qualified clinical study team member (e.g. MD, NP, PA, CDE) will assess and discuss the transition back to usual care with the study participant. |
| 673<br>674<br>675 | Participants will be asked to continue monitoring ketone levels for 24-48 hours after the hotel admission if ketones were >0.6 mmol/L prior to discharge. Urine ketone supplies may be provided for this testing. |
| 676<br>677<br>678 | All study equipment will be returned at the time of study end. Per investigator discretion, a participant may wear home the study CGM device in use and will be requested to return the study transmitter. |
| 679 | 7.9 Visit 5: Post Admission Check-In Visit |
| 680<br>681 | Approximately 24-48 hours after the hotel admission, the study team will contact the participant via phone/email/text to assess adverse events, adverse device effects, and device issues. |
| 682 | 7.10 Medical Monitor Review |
| 683<br>684 | At the conclusion of the Main Study, the medical monitor will review the data as referenced in section 8.3. |

Rocket-BPS 06-Oct-2022 

# **Chapter 8 Medical Monitor Review**

#### 8.1 Medical Monitor Study Safety Data Review

- The Medical Monitor will be provided all adverse event data for review to assess safety. The Medical Monitor will review data related to individual stopping criteria as detailed in the study
- 689 protocol.

685

686

690

#### 8.2 Medical Monitor Main Study Safety Data Review

- A Medical Monitor will review compiled safety data at the conclusion of the trial. In addition, the Medical Monitor will review all DKA and severe hypoglycemia irrespective of relatedness to study device use, and all serious events (including UADEs) related to study device use at the time of occurrence. The Medical Monitor also will be informed of any ADEs not meeting criteria for a UADE if the Study PI requests the Medical Monitor review. The Medical Monitor can request modifications to the study protocol or suspension or stoppage of the study if deemed necessary
- based on the totality of safety data available.

Rocket-BPS 06-Oct-2022 

| Chapter 9 Testing Procedures |
|---|
| 9.1 Laboratory / Point of Care Testing |
| 9.1.1 HbA1c |
| A blood sample will be obtained at screening to obtain a baseline hemoglobin A1c level. A blood test obtained within 2 weeks prior to enrollment may be used. |
| HbA1c level may be measured by study team using the DCA2000, a comparable point of care device, at time of screening |
| Labs may be obtained at a local laboratory (e.g. LabCorp) convenient to the participant. |
| 9.1.2 Pregnancy Test |
| A serum or urine pregnancy test will be required for women of childbearing potential at in person visit and admission. Test must be negative to participate in the study. |
| 9.1.3 Covid-19 Testing |
| All participants and study staff (e.g. on-site research coordinators, technicians, nurses, and physicians) will be tested with a COVID-19 test within the first 24 hours of the hotel admission or up to 72 hours in advance of being on-site for the Pilot and Main Study. Individuals with Covid-19 positive tests will be excluded from the study. |
| 9.1.4 Demographic Data Survey |
| The Demographic Date Survey will be asked often study eligibility has been mot |

The Demographic Data Survey will be asked after study eligibility has been met.
# **Chapter 10 Risks Associated with Clinical Trial**

#### 10.1 Potential Risks and Benefits of the Investigational Device

- Risks and Benefits are detailed below. Loss of confidentiality is a potential risk; however, data are handled to minimize this risk. Hypoglycemia, hyperglycemia and ketone formation are always a
- risk in participants with type 1 diabetes and participants will be monitored for these symptoms.

### 10.1.1 Venipuncture Risks

- A hollow needle/plastic tube may be placed in the arm for taking blood samples (e.g. external
- 723 HbA1c measurements for inclusion criteria). Blood draws can cause some common reactions like
- pain, bruising, or redness at the sampling site. Less common reactions include bleeding from the
- sampling site, formation of a small blood clot or swelling of the vein and surrounding tissues, and
- 726 fainting.

716

717

721

727

743

#### 10.1.2 Fingerstick Risks

- About 1 drop of blood will be removed by fingerstick for measuring blood sugars and sometimes
- HbA1c or other tests. This is a standard method used to obtain blood for routine hospital laboratory
- 730 tests. Pain is common at the time of lancing. In about 1 in 10 cases, a small amount of bleeding
- under the skin will produce a bruise. A small scar may persist for several weeks. The risk of local
- infection is less than 1 in 1000. This should not be a significant contributor to risks in this study
- as finger sticks are part of the usual care for people with diabetes.

#### 734 **10.1.3 Subcutaneous Catheter Risks (CGM)**

- Participants using the CGM will be at low risk for developing a local skin infection at the site of
- the sensor needle placement. If a catheter is left under the skin for more than 24 hours it is possible
- 737 to get an infection where it goes into the skin, with swelling, redness and pain. There may be
- bleeding where the catheter is put in and bleeding under the skin causes a bruise (1 in 10 risk).
- 739 Study staff should verbally alert the participant that on rare occasions, the CGM may break and
- leave a small portion of the sensor under the skin that may cause redness, swelling, or pain at the
- 741 insertion site. The participant should be further instructed to notify the study coordinator
- 742 immediately if this occurs.

#### 10.1.4 Risks of Hypoglycemia

- As with any person having type 1 diabetes and using insulin, there is always a risk of having a low
- blood sugar (hypoglycemia). The frequency of hypoglycemia should be no more and possibly less
- 746 than it would be as part of daily living. Symptoms of hypoglycemia can include sweating,
- 747 jitteriness, and not feeling well. Just as at home, there is the possibility of fainting or seizures
- 748 (convulsions) and that for a few days the participant may not be as aware of symptoms of

Rocket-BPS 06-Oct-2022 

hypoglycemia. A CGM functioning poorly and significantly over-reading glucose values could lead to inappropriate insulin delivery.

#### 10.1.5 Risks of Hyperglycemia

Hyperglycemia is likely because of the study design including unannounced carbohydrate ingestion. Also, hyperglycemia and ketonemia could occur if insulin delivery is attenuated or suspended for an extended period or if the pump or infusion set is not working properly. A CGM functioning poorly and significantly under-reading glucose values could lead to inappropriate suspension of insulin delivery.

#### 10.1.6 Risks of Device Reuse

Participant will be informed that FDA or relevant national authorities have approved the insulin pump, CGM, glucometer and ketone meter for single use and that by using them among multiple patients, bloodborne pathogens (i.e. Hepatitis B) may be spread through the use of multiple users.

- The study CGM system is labelled for single use only. The sensor (the component of the system that enters the skin) will be single use only. The transmitter and receiver may be reused during the study after cleaning the device using a hospital-approved cleaning procedure. The transmitter is attached to the sensor but does not enter the skin and the receiver, if used, is a handheld device.
- The study insulin pumps are labelled for single-patient use. During the study, this device may be reused after cleaning adhering to a hospital-approved cleaning procedure. All infusion set equipment will be single patient use only (infusion set insertion kits, tubing, cartridges etc.).
- The study blood glucose meter and blood ketone meter are labelled for single-patient use.

  During the study, these devices may be reused after cleaning adhering to a hospital-approved cleaning procedure.

## **10.1.7 Device Cleaning Instructions**

CGM cleaning instructions are provided in the Dexcom G4 Platinum (Professional) Cleaning and Disinfection manual (current edition) and a similar approach will be applied for the G6 version used in this study. The transmitter should be cleaned with Clorox Healthcare® Bleach Germicidal Cleaner or any disinfectant product in a spray bottle containing a bleach solution of 6500 parts per million with the EPA registration number 56392-7. The transmitter will be submerged in this solution and then placed on an absorbent wipe or clean surface. Two sprays will be dispensed from the Clorox cleaner onto each side of the transmitter. A nylon brush will be used to scrub the transmitter on all sides for 30 seconds. The transmitter will be placed in the Clorox Cleaner solution for one minute. Transmitter is then rinsed under flowing tap water for ten seconds. The transmitter will then be disinfected using a disinfectant product with EPA registration number 56392-7 using similar procedures as the cleaning process.

Rocket-BPS 06-Oct-2022 

- Per the pump manufacturer, the insulin pump will be cleaned with a damp lint-free cloth. Use of
- household or industrial cleaners, solvents, bleach, scouring pads, chemicals, or sharp instruments
- are prohibited. The pump should never be submerged in water. If needed, use only a very mild
- detergent, such as a bit of liquid soap with warm water. A soft towel will be used to dry the pump.
- 787 The glucometer is cleaned and disinfected with two separate Super Sani-Cloths (EPA number
- 788 9480-4). The entire surface will be cleaned, making sure the surface stays wet for 2 minutes. This
- step is repeated with a clean cloth for disinfecting the device.
- 790 The Precision Xtra User's Guide suggests that healthcare professionals use 10% bleach, 70%
- alcohol or 10% ammonia to clean the device.
- 792 Equipment that touches intact skin will be cleaned with ethyl or isopropyl alcohol (70-90%),
- 793 quaternary ammonium germicidal detergent (i.e. Cavicide, EPA number 46781) or household
- bleach. The contact time on the surface depends on the method used to clean the equipment.
- 795 Cavicide requires three minutes on the surface of the equipment. Clorox Germicidal Bleach Wipes
- require two minutes on the equipment. The surface should remain wet (i.e. slightly damp) with the
- disinfectant to be considered effective though not wet enough to leave drops of liquid.
- 798 In the event a manufacturer updates cleaning procedures for their device, the study team will
- adhere to the most current recommendations.
- 800 There is the risk of blood sampling collection and contamination from sampling techniques. Hand
- washing with either soap & water or waterless hand sanitizer will be used prior to caring for the
- study subject. Gloves will be worn during blood sample collection and processing. Medical
- personnel will continue to practice hygiene for the subject's protection (i.e. hand washing,
- 804 changing gloves frequently, disposing needles properly). Gloves will be removed, and hands
- washed or sanitized prior to leaving and upon return to the subject's room. Soiled linen will be
- changed to minimize the transfer of pathogenic organisms.

#### 10.1.8 Risk of Exercise

- There is a risk of musculoskeletal symptoms or injury from participating in an exercise regimen.
- 809 There are cardiovascular or cerebrovascular risks (including but not limited to dizziness,
- 810 lightheaded, syncope, arrhythmia or ischemia) associated with participating in an exercise
- regimen. The intention of the eligibility criteria will be to minimize these risks.

#### 812 **10.1.9 Hb1Ac Risk**

807

813 An NGSP Point of Care analyzer (i.e. DCA Vantage Analyzer) will be utilized at the research site

814 to obtain the subject's HbA1c level.

Rocket-BPS 06-Oct-2022 

| 815 | 10.1.10 Other Risks |
|---|---|
| 816<br>817<br>818<br>819<br>820 | Some participants may develop skin irritation or allergic reactions to the adhesives used to secure the CGM, or to secure the insulin infusion sets for the continuous subcutaneous insulin infusion. If these reactions occur, different adhesives or "under-taping" (such as with IV 3000, Tegaderm etc.) will be tried, sites will be rotated frequently, and a mild topical steroid cream or other medication may be required. |
| 821<br>822<br>823<br>824<br>825<br>826 | Whenever the skin is broken there is the possibility of an infection. The CGM and pump infusion sites are inserted under the skin. It is possible that any part that is inserted under the skin may cause an infection. These occur very infrequently, but, if an infection was to occur, oral and/or topical antibiotics can be used. The risk of skin problems could be greater if you use a sensor for longer than it is supposed to be used. Therefore, participants will be carefully instructed about proper use of the sensor. |
| 827<br>828<br>829 | Data downloaded from the CGM, pump, glucometer, and ketone meter will be collected for the study as measures of diabetes self-management behaviours. Some people may be uncomfortable with the researchers' having such detailed information about their daily diabetes habits. |
| 830 | 10.1.11 Known Potential Benefits |
| 831<br>832<br>833 | It is expected that this protocol will yield increased knowledge about using an automated closed-loop system with anticipatory action to control glucose levels. The individual participant may no benefit from study participation. |
| 834 | 10.1.12 Risk Assessment |
| 835<br>836<br>837<br>838<br>839<br>840<br>841<br>842<br>843 | Based on the facts that (1) adults with diabetes experience mild hypoglycemia and hyperglycemia frequently as a consequence of the disease and its management, (2) the study intervention involves periodic automated insulin dosing that may increase the likelihood of hypoglycemia, and periodic automated attenuation of insulin delivery that may increase the likelihood of hyperglycemia, (3) mitigations are in place, and have been tested in prior studies using the investigational device system in the home setting, that limit the likelihood of excessive insulin dosing or prolonged withdrawal of insulin, and (4) rapid reversal of hypoglycemia and hyperglycemia can be achieved. In addition, it is the belief of the investigators that this study also presents prospect of direct benefit to the participants and general benefit to others with diabetes. |
| 844 | 10.2 General Considerations |
| 845<br>846<br>847 | The study is being conducted in compliance with the policies described in the study policies document, with the ethical principles that have their origin in the Declaration of Helsinki, with the protocol described herein, and with the standards of Good Clinical Practice (GCP). |
| 848<br>849 | Whenever possible, data will be directly collected in electronic case report forms, which will be considered the source data. |

Rocket-BPS 06-Oct-2022 

853

854

855

856

857

858

859

860

861

862

863

864

865

866

867

| 850 | The protocol is considered a significant risk device study, due to the fact that the closed-loop |
|---|---|
| 851 | system is experimental. Therefore, an investigational device exemption (IDE) from the U.S. Food |
| 852 | and Drug Administration (FDA) is required to conduct the study. |

#### 10.3 COVID-19 Risk Mitigation Plan and Justification

The study team will follow local guidelines that are in effect at the time of the study admission.

#### 10.3.1 Participants and Study Personnel

We will follow a combination of approaches to increase our likelihood of having a COVID-free environment:

- We will follow CDC and local guidelines in effect at the time of the study.
- All participants and study staff (research coordinators, technicians, nurses, and physicians) will be tested with an FDA authorized COVID-19 test with the **first 24 hours of study start or up to approximately 72 hours before their participation in the study hotel**. Those with positive tests will be excluded from the study.
- Any participants with positive test will be discharged from the study. Hotel rooms of these participants will be restricted from future use. We will limit any personal interaction between study personnel and these individuals. We will follow local guidelines in effect at the time of study to guide interactions.

#### 10.3.2 Environment

The study team will adhere to current hotel guidelines.

Rocket-BPS 06-Oct-2022 

899

900

901

#### Chapter 11 Adverse Events, Device Issues, and Stopping Rules 869 11.1 Definitions 870 871 11.1.1 Adverse Events (AE) 872 Any untoward medical occurrence in a study participant, irrespective of the relationship between the adverse event and the device(s) under investigation (section 11.2) for reportable adverse events 873 874 for this protocol). 875 Positive pregnancy test will be not considered adverse event. 876 11.1.2 Serious Adverse Event (SAE) 877 Any untoward medical occurrence that: 878 • Results in death. 879 • Is life-threatening; (a non-life-threatening event which, had it been more severe, might 880 have become life-threatening, is not necessarily considered a serious adverse event). • Requires inpatient hospitalization or prolongation of existing hospitalization. 881 882 • Results in persistent or significant disability/incapacity or substantial disruption of the 883 ability to conduct normal life functions (life threatening). 884 • Is a congenital anomaly or birth defect. • Is considered a significant medical event by the investigator based on medical judgment 885 886 (e.g., may jeopardize the participant or may require medical/surgical intervention to 887 prevent one of the outcomes listed above). 888 11.1.3 Unanticipated Adverse Device Effect (UADE) 889 Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, 890 891 severity, or degree of incidence in the investigational plan or application (including a 892 supplementary plan or application), or any other unanticipated serious problem associated with a 893 device that relates to the rights, safety, or welfare of participants (21 CFR 812.3(s)). 894 11.1.4 Adverse Device Effect (ADE) 895 Any untoward medical occurrence in a study participant which the device may have caused or to 896 which the device may have contributed. 897 11.1.5 Device Complaints and Malfunctions 898 A device complication or complaint is something that happens to a device or related to device

Rocket-BPS 06-Oct-2022 

performance, whereas an adverse event happens to a participant. A device complaint may occur

independently from an AE, or along with an AE. An AE may occur without a device complaint or

there may be an AE related to a device complaint. A device malfunction is any failure of a device

to meet its performance specifications or otherwise perform as intended. Performance specifications include all claims made in the labelling for the device. The intended performance of a device refers to the intended use for which the device is labelled or marketed. (21 CFR 803.3).

#### 11.2 Reportable Events

For this protocol, a reportable adverse event includes any untoward medical occurrence that meets one of the following criteria:

- A serious adverse event as defined in section 11.2
- An Adverse Device Effect as defined in section 11.1.4, unless excluded from reporting in section 11.7
- An Adverse Event as defined in section 11.1.1 occurring in association with a study procedure
- An AE as defined in section 11.1.1 which leads to discontinuation of a study device for 2 or more hours
- Hypoglycemia meeting the definition of severe hypoglycemia as defined in section 11.2.1
- Diabetic ketoacidosis (DKA) as defined in section 11.2.2 or in the absence of DKA, a hyperglycemic or ketosis event meeting the criteria defined below

Hypoglycemia and hyperglycemia not meeting the criteria below will not be recorded as adverse events unless associated with an Adverse Device Effect. Skin reactions from sensor placement are only reportable if severe and/or required treatment.

#### 11.2.1 Hypoglycemia Event

- Hypoglycemia not associated with an Adverse Device Effect is only reportable as an adverse event when the following definition for severe hypoglycemia is met:
  - The event required assistance of another person due to altered consciousness, and required another person to actively administer carbohydrate, glucagon, or other resuscitative actions
  - Impaired cognitively to the point that he/she was unable to treat himself/herself, was unable to verbalize his/ her needs, was incoherent, disoriented, and/or combative, or experienced seizure or coma. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma
  - If plasma glucose measurements are not available during such an event, neurological recovery attributable to the restoration of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration

## 11.2.2 Hyperglycemia Events/Diabetes Ketoacidosis

- Hyperglycemia not associated with an Adverse Device Effect is only reportable as an adverse event when one of the following four criteria is met:
  - The event involved DKA, as defined by the Diabetes Control and Complications Trial (DCCT) and described below evaluation or treatment was obtained at a health care provider facility for an acute event involving hyperglycemia or ketosis

Rocket-BPS 06-Oct-2022 

941

942

944

945

946

952

958

959

960

961

962

963

964 965

966

967

968

- Blood ketone level ≥1.5 mmol/L and communication occurred with a health care provider at the time of the event
  - Blood ketone level ≥3.0 mmol/L, even if there was no communication with a health care provider
- 943 Hyperglycemic events are classified as DKA if the following are present:
  - Symptoms such as polyuria, polydipsia, nausea, or vomiting
  - Serum ketones >1.5 mmol/L or large/moderate urine ketones
  - Either arterial blood pH <7.30 or venous pH <7.24 or serum bicarbonate <15
- Treatment provided in a health care facility
- All reportable Adverse Events—whether volunteered by the participant, discovered by study personnel during questioning, or detected through physical examination, laboratory test, or other means—will be reported on an adverse event form online. Each adverse event form is reviewed by the Medical Monitor to verify the coding and the reporting that is required.

#### 11.3 Relationship of Adverse Event to Study Device

- The study investigator will assess the relationship of any adverse event to be related or unrelated by determining if there is a reasonable possibility that the adverse event may have been caused by the study device.
- To ensure consistency of adverse event causality assessments, investigators should apply the following general guideline when determining whether an adverse event is related:
  - There is a plausible temporal relationship between the onset of the adverse event and the study intervention, and the adverse event cannot be readily explained by the participant's clinical state, intercurrent illness, or concomitant therapies; and/or the adverse event follows a known pattern of response to the study intervention; and/or the adverse event abates or resolves upon discontinuation of the study intervention or dose reduction and, if applicable, reappears upon rechallenge.
  - Evidence exists that the adverse event has an etiology other than the study intervention (e.g., pre-existing medical condition, underlying disease, intercurrent illness, or concomitant medication); and/or the adverse event has no plausible temporal relationship to study intervention.

#### 11.4 COVID-19 Transmission

- While we are taking steps to prevent transmission of COVID-19 during this study, there is a possibility that participants, based either on exposure before the hotel admission or during the stay,
- are infected with COVID-19. Any appearance of significant COVID-19 symptoms in participants
- will be cause for repeat COVID-19 testing and possible quarantine until test results are returned.
- 973 If this Covid-19 test is positive, the participant will be discharged from the study.
- 974 In the event of a COVID-19 positive test in a participant, the study team will follow up with the
- participant via phone until conclusion of treatment for the COVID-19 related symptoms. All

Rocket-BPS 06-Oct-2022 

participants will be asked to follow up via phone with the study team in the event of a positive test within 14 days after discharge from the hotel.

#### 11.5 Intensity of Adverse Event

- The intensity of an adverse event will be rated on a three-point scale: (1) mild, (2) moderate, or (3) severe. It is emphasized that the term severe is a measure of intensity: thus, a severe adverse event is not necessarily serious. For example, itching for several days may be rated as severe, but may not be clinically serious.
  - MILD: Usually transient, requires no special treatment, and does not interfere with the participant's daily activities.
  - MODERATE: Usually causes a low level of inconvenience or concern to the participant and may interfere with daily activities but is usually ameliorated by simple therapeutic measures.
  - SEVERE: Interrupts a participant's usual daily activities and generally requires systemic drug therapy or other treatment.

### 11.6 Coding of Adverse Events

- Adverse events will be coded per the UVA IRB website instructions (i.e. mild, moderate, severe).
- The Medical Monitor will review the investigator's assessment of causality and may agree or
- 993 disagree. Both the investigators and Medical Monitor's assessments will be recorded. The
- Medical Monitor will have the final say in determining the causality.
- Adverse events that continue after the participant's discontinuation or completion of the study will
- be followed until their medical outcome is determined or until no further change in the condition
- 997 is expected.

978

983

984

985

986

987

988 989

990

998

1002

1003

1004

1005

1006

1007

1008 1009

1010

1011

#### 11.7 Outcome of Adverse Events

- The outcome of each reportable adverse event will be classified by the investigator as follows:
- RECOVERED/RESOLVED The participant recovered from the AE/SAE without sequelae. Record the AE/SAE stop date.
  - RECOVERED/RESOLVED WITH SEQUELAE The event persisted and had stabilized without change in the event anticipated. Record the AE/SAE stop date.
  - FATAL A fatal outcome is defined as the SAE that resulted in death. Only the event that was the cause of death should be reported as fatal. AEs/SAEs that were ongoing at the time of death; however, were not the cause of death, will be recorded as "resolved" at the time of death.
  - NOT RECOVERED/NOT RESOLVED (ONGOING) An ongoing AE/SAE is defined as the event was ongoing with an undetermined outcome.
  - An ongoing outcome will require follow-up by the site in order to determine the final outcome of the AE/SAE.

Rocket-BPS 06-Oct-2022 

1014

1015

1016

1017

1018 1019

1020

1026

1031

1032

1033

1035

1036

1037 1038

1039

1040

1041 1042

1043

1044

1045 1046

1047 1048

- The outcome of an ongoing event at the time of death that was not the cause of death, will be updated and recorded as "resolved" with the date of death recorded as the stop date.
  - UNKNOWN An unknown outcome is defined as an inability to access the participant or the participant's records to determine the outcome (for example, a participant that was lost to follow-up).
  - All clinically significant abnormalities of clinical laboratory measurements or adverse events occurring during the study and continuing at study termination should be followed by the participant's physician and evaluated with additional tests (if necessary) until diagnosis of the underlying cause, or resolution. Follow-up information should be recorded on source documents.
- If any reported adverse events are present when a participant completes the study, or if a participant is withdrawn from the study due to an adverse event, the participant will be contacted for reevaluation within 2 weeks. If the adverse event has not resolved, additional follow-up will be performed as appropriate. Every effort should be made by the Investigator or delegate to contact the participant until the adverse event has resolved or stabilized.

### 11.8 Reportable Device Issues

- All UADEs, ADEs, device complaints, and device malfunctions will be reported irrespective of whether an adverse event occurred, except in the following circumstances.
- The following device issues are anticipated and will not be reported but will reported as an Adverse Event if the criteria for AE reporting described above are met:
  - Component disconnections
    - CGM sensors lasting fewer than the number of days expected per CGM labelling
  - CGM tape adherence issues
- Pump infusion set occlusion not leading to ketosis
  - Battery lifespan deficiency due to inadequate charging or extensive wireless communication
    - Intermittent device component disconnections/communication failures not leading to system replacement
    - Device issues clearly addressed in the user guide manual that do not require additional troubleshooting
    - Skin reactions from CGM sensor placement or pump infusion set placement that do not meet criteria for AE reporting

#### 11.9 Timing of Event Reporting

- UADEs must be reported within 10 working days to the FDA after the sponsor first receives notice of the adverse effect.
- Other reportable adverse events, device malfunctions (with or without an adverse event) and device complaints should be reported promptly, but there is no formal required reporting period.

Rocket-BPS 06-Oct-2022 

1052 1053

1054

1055 1056

1057 1058

1059

1060

1061

1062

1063

1064 1065

1066

1067

1068 1069

1070

1071

1072

- The IDE Sponsor will investigate the UADE and if indicated, report the results of the investigation to the IRBs, FDA, and DSMB within 10 working days of the study team becoming aware of the UADE per 21CFR 812.46(b) (2).
  - The Medical Monitor will determine if the UADE presents an unreasonable risk to participants. If so, the DSMB must ensure that all investigations, or parts of investigations presenting that risk, are terminated as soon as possible but no later than 5 working days after the Medical Monitor makes this determination and no later than 15 working days after first receipt notice of the UADE.
  - In the case of a device system component malfunction (e.g. pump, CGM, control algorithm), information will be forwarded to the responsible manufacturer by the study personnel.

### 11.10 Stopping Criteria

# 11.10.1 Participant Discontinuation

Rules for discontinuing study device use are described below.

- The investigator believes it is unsafe for the participant to continue the intervention. This could be due to the development of a new medical condition or worsening of an existing condition; or participant behaviour contrary to the indications for use of the device that imposes on the participant's safety
- The participant requests that the treatment be stopped
- The participant tests positive for COVID-19 (during study testing or otherwise within 14 days of study start) or subsequently develops symptoms for COVID-19 and tests positive.
- Diagnosis of DKA. Any severe hypoglycemia event meeting the definition in section 11.2.1 of the protocol.

#### 11.10.2 Suspending/Stopping Overall Study

- In the case of an unanticipated system malfunction resulting in a severe hypoglycemia or severe hyperglycemia event (as defined in section 11.2.2), use of the study device system will be suspended while the problem is diagnosed.
- In the event that two distinct episodes of DKA or two distinct severe hypoglycemia events as defined in section 11.2 occur, the overall study would be suspended while the underlying conditions are determined.
- In addition, study activities could be similarly suspended if the manufacturer of any constituent study device requires stoppage of device use for safety reasons (e.g. product recall). The affected study activities may resume if the underlying problem can be corrected by a protocol or system modification that will not invalidate the results obtained prior to suspension. The study Medical Monitor will review all adverse events and adverse device events that are reported during the study and will review compiled safety data at periodic intervals. The Medical Monitor may request suspension of study activities or stoppage of the study if deemed necessary based on the totality

1086 of safety data available.

| 1087 | 11.11 Independent Safety Oversight |
|---|---|
| 1088 | A Medical Monitor will review all DKA and severe hypoglycemia irrespective of relatedness to |
| 1089 | study device use, and all serious events (including UADEs) related to study device use at the time |
| 1090 | of occurrence. The Medical Monitor can request modifications to the study protocol or suspension |
| 1091 | or outright stoppage of the study if deemed necessary based on the totality of safety data available. |
| 1092 | Details regarding Medical Monitor review will be documented in a separate Medical Monitor |
| 1093 | document. |
| 1094 | 11.12 Definition of a Data Breach |
| 1095 | A data breach is defined in the HITECH Act (43 USC 17932) as an unauthorized acquisition, |
| 1096 | access, or use of protected health information (PHI) that compromises the security or privacy of |
| 1097 | such information. |

Rocket-BPS 06-Oct-2022 

1098

1112

**Chapter 12 Miscellaneous Considerations** 

#### 1099 12.1 Prohibited Medications, Treatments, and Procedures 1100 Participants using glulisine at the time of enrollment will be asked to contact their personal physician to change their prescribed personal insulin to lispro or aspart for the duration of the trial. 1101 1102 The study devices (study insulin pump, study CGM) must be removed before Magnetic Resonance 1103 Imaging (MRI), Computed Tomography (CT) or diathermy treatment. Participants may continue 1104 in the trial after temporarily discontinuing use if requiring one of the treatments above. 1105 12.2 Participant Withdrawal 1106 Participation in the study is voluntary. Participant may withdraw at any time. For participants who 1107 do withdraw from the study, the study team will determine if their data will be used in analysis. 1108 12.3 Confidentiality For security and confidentiality purposes, subjects will be assigned an identifier that will be used 1109 instead of their name. Protected health information gathered for this study may be shared with the 1110 1111 third-party collaborators. De-identified subject information may also be provided to collaborators

involved in the study after the appropriate research agreement has been executed.

1113

1143

| 1113 | <b>Chapter 13 Statistical Consideration</b> |
|---|---|
| 1114 | 13.1 Design and Randomization |
| 1115<br>1116 | The main study is itself an early exploratory study to assess glycemic responses of a fully closed-loop system (Rocket AP). This information is detailed in Table 1. |
| 1117 | Randomization will occur via selection from the above list using permuted blocks in groups of 4. |
| 1118 | 13.1.1 Planned Analysis |
| 1119<br>1120 | Our primary objective is to assess the impact of priming bolus on post prandial FCL control therefore we will test the following statistical hypotheses |
| 1121 | |
| 1122<br>1123 | a. Null Hypothesis: There is no difference in the means of time spent in the 70-180mg/dL range during daytime between FCL with and without prandial priming bolus (BPS at 6% and 0% of TDI respectively) |
| 1124 | |
| 1125<br>1126 | b. Alternative Hypothesis: There is a difference in the means of time spent in the 70-180mg/dL range during daytime between FCL with and without prandial priming bolus (BPS at 6% and 0% of TDI respectively) |
| 1127 | |
| 1128<br>1129 | To do so we will use repeated measure ANOVA models to predict daytime time in range with the BPS status a fixed effect and baseline HbA1c and gender as covariates. |
| 1130 | |
| 1131 | Secondary outcomes: |
| 1132<br>1133<br>1134<br>1135<br>1136 | All secondary outcomes will be similarly analyzed. If an outcomes distribution is not suited for mixed model analysis (e.g. profound skewness, or large atom at boundary) we will perform paired Wilcoxon signed rank test (and loose the capacity to use covariate) to test difference in the median instead of the mean; this is expected for time below 70mg/dL, number of hypoglycemia, and possibly time above 250mg/dL. |
| 1137 | |
| 1138 | We do not plan to correct for multiple comparisons. |
| 1139 | |
| 1140<br>1141<br>1142 | We do not expect substantial missing values in this highly supervised study, but if more than 3 subjects have one or more missing admissions, we will consider switching from RANOVA to mixed model repeated measures. |

| 13.2 Sample Size |
|---|
| a early exploratory Study, the goal will be to complete up to 20 participants in the main study provide data from a variety of individuals. This number was chosen out of feasibility and no ma formal power calculation. (The Pilot Study for this proposal will assess ease of system and be completed in a minimum of 2-3 individuals prior to the beginning of the Main Study.) With 20 and our randomized crossover design (allowing for paired comparison), we can hope to detect a imum effect size of 0.66 at a power of 80%. Based of prior FCL study, the standard deviation of daytime is approximately 12%, leading to a detectable difference in daytime TIR of 8%. |
| 13.3 Outcome Measures |
| 13.3.1 Primary Efficacy Endpoint |
| e study design allows for multiple comparisons of blood glucose control during the study meals exercise sessions, with for the primary comparison of interest being between the RocketAF and without BPS. Our primary endpoint is CGM time-in-range 70-180 mg/dL for the daytime and $6 \text{ am} - 12 \text{ am}$ when on each treatment modality (BPS vs. no BPS). |
| 13.3.2 Secondary Outcomes |
| h admission is separated into windows of analysis: |
| <ul> <li>The entirety of the admission (24h: 4pm to 4pm)</li> <li>The 4 hours following each of the meals.</li> <li>The overnight period (12 am to 6 am)</li> </ul> |
| each of these periods we will compute the following outcomes: |
| <ul> <li>Number of hypoglycemia events defined as at least two consecutive CGM values &lt;70mg/dL or a hypoglycemia treatment (two events separated by less than 30 minutes are counted as one).</li> <li>Percent CGM time &lt;70 mg/dL</li> <li>Percent CGM time between 80-140mg/dL</li> <li>Percent CGM time between 70-180mg/dL</li> <li>Percent CGM time &gt;180 mg/dL</li> <li>Percent CGM time &gt;250 mg/dL</li> <li>Units of insulin injected</li> <li>Area under the curve when accounting for starting BG</li> <li>Low Blood Glucose Index</li> <li>High Blood Glucose Index</li> <li>CGM coefficient of variation</li> <li>Mean CGM</li> </ul> |

| 1179 | 13.3.3 CGM data treatment |
|---|---|
| 1180<br>1181 | • Saturated CGM values "High" and "Low" will be replaced by 401mg/dL and 39mg/dL respectively. |
| 1182<br>1183<br>1184<br>1185<br>1186 | <ul> <li>Any CGM gaps shorter than 1 hour will be interpolated</li> <li>CGM data during recorded occlusion event will be removed from analysis as follow: any measurement less than 2h before or after the time of record will be removed.</li> <li>CGM data following a pump/DiAs communication interruption &gt;1h by less than 2h will be removed</li> </ul> |
| 1187 | 13.3.4 Outcome computation conditions |
| 1188<br>1189 | Outcomes will only be computed if at least 80% of the analysis window CGM measurements (after data treatment) are available |
| 1190 | 13.4 Safety Analyses |
| 1191<br>1192<br>1193 | We will assess for the system's functionality, including the ability of the system to run its code without error (delivering insulin safely, as planned), as well as its ability to avoid low BG <70 mg/dL. |
| 1194 | 13.5 Baseline Descriptive Statistics |
| 1195<br>1196<br>1197 | Baseline demographic and clinical characteristics of the cohort of all randomized participants will be summarized in a table using summary statistics appropriate to the distribution of each variable. Descriptive statistics will be displayed overall and by treatment group. |
| 1198 | Will include: |
| 1199<br>1200<br>1201<br>1202<br>1203<br>1204<br>1205<br>1206<br>1207 | <ul> <li>Age</li> <li>HbA1c</li> <li>Gender</li> <li>Race/ethnicity</li> <li>CGM use before enrollment</li> <li>AID use before enrollment</li> <li>Diabetes duration</li> <li>BMI</li> <li>Total Daily Insulin</li> </ul> |
| 1208 | 13.6 Device Issues |
| 1209<br>1210 | The following tabulations and analyses will be performed during time on the UVa AP systems to assess device issues: |
| 1211<br>1212<br>1213 | <ul> <li>Device malfunctions requiring study team contact and other reported device issues</li> <li>% time CGM data available</li> <li>% time with closed loop control</li> </ul> |

1214

1215

1222

# **Chapter 14 Data Collection and Monitoring**

#### 14.1 Case Report Forms and Device Data

- 1216 The study data are collected through a combination of case report forms (electronic and paper) and
- 1217 electronic device data files obtained from the software and individual hardware components. These
- electronic device files and electronic CRFs are considered the primary source documentation.
- When data are directly collected in electronic case report forms, this will be considered the source
- data. Records will be maintained in accordance with ICH E6 and institutional regulatory
- requirements for the protection of confidentiality of participants.

# 14.2 Study Records Retention

- 1223 Study documents should be retained for a minimum of 2 years after the last approval of a marketing
- application in an ICH region and until there are no pending or contemplated marketing applications
- in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical
- development of the investigational product. These documents should be retained for a longer
- period, however, if required by local regulations. No records will be destroyed without the written
- consent of the sponsor, if applicable. It is the responsibility of the sponsor to inform the investigator
- when these documents no longer need to be retained.

#### 1230 **14.3 Protocol Deviations**

- 1231 A protocol deviation is any noncompliance with the clinical trial protocol, Good Clinical Practices
- 1232 (GCP), or procedure requirements. The noncompliance may be either on the part of the participant,
- the investigator, or the study site staff. As a result of deviations, corrective actions may be
- developed by the site and implemented as appropriate. Major deviations will be reported to the
- 1235 IRB-HSR within 7 calendar days of when the study team becomes aware of the event.

Rocket-BPS 06-Oct-2022 

# **Chapter 15 Ethics/Protection of Human Participants**

#### 15.1 Ethics Standard

1236

1237

1241

1248

1249

1250

- The investigator will ensure that this study is conducted in full conformity with Regulations for
- the Protection of Human Participants of Research codified in 45 CFR Part 46, 21 CFR Part 50, 21
- 1240 CFR Part 56, and/or the ICH E6.

#### 15.2 Institutional Review Boards

- The protocol, informed consent form(s), recruitment materials, and all participant materials will
- be submitted to the IRB for review and approval. Approval of both the protocol and the consent
- form must be obtained before any participant is enrolled. Any amendment to the protocol will
- require review and approval by the IRB before the changes are implemented to the study. All
- changes to the consent form will be IRB approved; a determination will be made regarding whether
- previously consented participants need to be re-consented.

#### 15.3 Informed Consent Process

#### 15.3.1 Consent Procedures and Documentation

- Informed consent is a process that is initiated prior to an individual's agreement to participate in
- the study and continues throughout the individual's study participation. Extensive discussion of
- risks and possible benefits of participation will be provided. Consent forms will be IRB approved
- and the participant will be asked to read and review the document. The investigator or their
- delegate will explain the research study to the participant and answer any questions that may arise.
- All participants will receive a verbal explanation in terms suited to their comprehension of the
- purposes, procedures, and potential risks of the study and of their rights as research participants.
- Participant will have the opportunity to carefully review the written consent form and ask questions
- 1258 prior to signing.
- The consenting process will involve discussing the study at length in a phone call/HIPAA
- compliant telecommunication method for consenting that is not face to face. The participant will
- sign the informed consent document prior to any procedures being done specifically for the study.
- The consent form may be signed electronically with the use of the Part 11 compliant version of
- DocuSign for both in-person and telecommunication screening visits. The study team will follow
- the FDA part 11 compliant process of verification of reviewing two forms of identification if
- signing electronically off site. A HIPAA compliant video conferencing tool will be utilized during
- 1266 the consenting process of the telecommunication screening visit to facilitate review of the
- 1267 participant's identification. A copy of the informed consent document will be given to the
- participant for their records. The rights and welfare of the participants will be protected by

Rocket-BPS 06-Oct-2022 

1289

emphasizing to them that the quality of their medical care will not be adversely affected if they 1269 decline to participate in this study. 1270 1271 15.3.2 Participant and Data Confidentiality 1272 The study monitor, representatives of the IRB or device company supplying study product may 1273 inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) for the participants in this study. 1274 1275 The study participant's contact information will be securely stored at the clinical site for internal 1276 use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by local IRB and Institutional regulations. 1277 1278 15.3.3 Participant and Data Confidentiality 1279 The study monitor, representatives of the IRB or device company supplying study product may inspect all documents and records required to be maintained by the investigator, including but not 1280 1281 limited to, medical records (office, clinic, or hospital) for the participants in this study. 1282 The study participant's contact information will be securely stored at the clinical site for internal 1283 use during the study. At the end of the study, all records will continue to be kept in a secure location 1284 for as long a period as dictated by local IRB and Institutional regulations. 1285 Study participant research data, which is for purposes of statistical analysis and scientific reporting, 1286 will be transmitted to and stored at the University of Virginia Center for Diabetes Technology. 1287 The study data entry and study management systems used by research staff will be secured and 1288 password protected. At the end of the study, all study databases may be de-identified and archived

at the University of Virginia Center for Diabetes Technology.

Rocket-BPS 06-Oct-2022 

# **Chapter 16 References**

- 1291 1. Burdick J, Chase HP, Slover RH, et al. Missed insulin meal boluses and elevated hemoglobin
- 1292 A(1c) levels in children receiving insulin pump therapy. Pediatrics. Mar 2004;113(3):E221-E224.
- 1293 doi:10.1542/peds.113.3.e221

1290

- 1294 2. Cherñavvsky DR, DeBoer MD, Keith-Hynes P, et al. Use of an artificial pancreas among
- adolescents for a missed snack bolus and an underestimated meal bolus. Pediatr Diabetes. Feb
- 1296 2016;17(1):28-35. doi:10.1111/pedi.12230
- 1297 3. Garcia-Tirado J, Brown SA, Laichuthai N, et al. Anticipation of Historical Exercise Patterns
- by a Novel Artificial Pancreas System Reduces Hypoglycemia During and After Moderate-
- 1299 Intensity Physical Activity in People with Type 1 Diabetes. Diabetes Technol Ther. Dec
- 1300 2020;doi:10.1089/dia.2020.0516
- 4. Voysey, Merryn and Costa Clemens, Sue Ann and Madhi, Shabir A. et al and Group, Oxford
- 1302 COVID Vaccine Trial, Single Dose Administration, And The Influence Of The Timing Of The
- Booster Dose On Immunogenicity and Efficacy Of ChAdOx1 nCoV-19 (AZD1222) Vaccine.
- 1304 Available at SSRN: https://ssrn.com/abstract=3777268